CLINICAL TRIAL: NCT01030965
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of GSK573719 Delivered Once-daily Over 28 Days in Subjects With COPD
Brief Title: 28-day Repeat Dose Study of GSK573719
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113589
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Bronchitis; Anticholinergic; Emphysema; Long-acting muscarinic antagonist; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK573719 125mcg (Experimental): 125mcg once-daily via novel dry powder inhaler
  Interventions: Drug: GSK573719 125mcg
- GSK573719 250mcg (Experimental): 250mcg once-daily via novel dry powder inhaler
  Interventions: Drug: GSK573719 250mcg
- GSK573719 500mcg (Experimental): 500mcg once-daily via novel dry powder inhaler
  Interventions: Drug: GSK573719 500mcg
- Placebo (Placebo Comparator): once-daily via novel dry powder inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK573719 125mcg — 125mcg once-daily
  Arms: GSK573719 125mcg
Drug: GSK573719 250mcg — 250mcg once-daily
  Arms: GSK573719 250mcg
Drug: GSK573719 500mcg — 500mcg once-daily
  Arms: GSK573719 500mcg
Drug: Placebo — once-daily
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy, safety, and pharmacokinetics of GSK573719 compared with placebo in subjects with COPD

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate 3 doses of GSK573719 administered once-daily over 28 days in subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent prior to study participation
* Males or females of non-childbearing potential
* 40 to 80 years of age
* COPD diagnosis
* 10 pack-years history or greater of cigarette smoking
* Post-bronchodilator FEV1/FVC ratio of 0.70 or less
* Post-bronchodilator FEV1 of 25 to 70% of predicted normal

Exclusion Criteria:

* Asthma
* Other significant respiratory disorders besides COPD, including alpha-1 deficiency
* Previous lung resection surgery
* Chest X-ray or CP scan showing clinically significant abnormalities not due to COPD
* Use of oral steroids or antibiotics for a COPD exacerbation within 6 weeks of screening
* Hospitalization for COPD or pneumonia within 3 months of screening
* Any significant disease that would put subject at risk through study participation
* BMI greater than 35
* Pacemaker
* Significantly abnormal ECG or clinical lab finding (including Hepatitis B or C)
* Cancer
* Allergy or hypersensitivity to anticholinergics or inhaler excipients
* Diseases that would contraindicate the use of anticholinergics
* Use of oral corticosteroids within 6 weeks of screening
* Use of long-acting beta-agonists within 48 hours of screening
* Use of tiotropium within 14 days of screening
* Use of theophyllines or anti-leukotrienes within 48 hours of screening
* Use of short-acting bronchodilators within 4 to 6 hours of screening
* Use of investigational medicines within 30 days of screening
* Use of high dose inhaled corticosteroids
* Use of long-term oxygen therapy, CPAP or NIPPV
* Participation in acute phase of pulmonary rehabilitation program
* History of alcohol or drug abuse within 2 years prior to screening
* History of psychiatric disease limiting validity of consent
* Affiliation with the investigative site
* Previous use of GSK573719

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2009-12-15 (Actual); Primary Completion 2010-07-04 (Actual); Study Completion 2010-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (4):
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (5):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gidle
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Decramer M, Maltais F, Feldman G, Brooks J, Harris S, Mehta R, Crater G. Bronchodilation of umeclidinium, a new long-acting muscarinic antagonist, in COPD patients. Respir Physiol Neurobiol. 2013 Jan 15;185(2):393-9. doi: 10.1016/j.resp.2012.08.022. Epub 2012 Sep 28. PMID 23026438
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113589 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a Run-in Period of 5 to 8 days, followed by a 28-day Treatment Period. A total of 421 participants were screened; of these, 125 were screen failures, 10 were Run-in failures, 288 were randomized, and 285 received at least one dose of study drug (three participants were randomized but did not receive study drug).
Groups:
- Placebo: Participants received matching placebo once daily (QD) in the morning via a dry powder inhaler (DPI) for 28 days.
- UMEC 125 µg: Participants received umeclidinium bromide (UMEC) 125 micrograms (µg) QD in the morning via a DPI for 28 days.
- UMEC 250 µg: Participants received UMEC 250 µg QD in the morning via a DPI for 28 days.
- UMEC 500 µg: Participants received UMEC 500 µg QD in the morning via a DPI for 28 days.
Period: Overall Study
Arm/Group | Placebo | UMEC 125 µg | UMEC 250 µg | UMEC 500 µg
Started | 71 | 71 | 72 | 71
Completed | 67 | 65 | 68 | 64
Not Completed | 4 | 6 | 4 | 7
Not completed — Lack of Efficacy | 3 | 2 | 0 | 3
Not completed — Protocol Violation | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 1
Not completed — Protocol-defined Stopping Criteria | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC 125 µg | UMEC 250 µg | UMEC 500 µg | Total
Number analyzed (Participants) | 71 | 71 | 72 | 71 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (6.80) | 60.1 (8.75) | 60.3 (8.45) | 62.6 (9.30) | 61.4 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 35 | 30 | 34 | 123
  Male | 47 | 36 | 42 | 37 | 162
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 4 | 3 | 1 | 9
  White | 70 | 67 | 69 | 69 | 275
  African American/African Heritage & White | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Day 29
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Treatment Day 29 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after dosing on Day 28. Baseline is defined as the mean of the FEV1 values obtained at 30 minutes and immediately pre-dose on Day 1. Change from Baseline is defined as the difference between trough on Day 29 and Baseline. Analysis was performed using a repeated measures model with covariates of Baseline (BL), country, sex, age, treatment, smoking status, day, day by Baseline interaction, and day by treatment interaction.
Time Frame: Baseline and Day 29
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received >=1 dose of randomized study medication in the treatment period. All participants with >=1 post-BL assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 29.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 125 µg | UMEC 250 µg | UMEC 500 µg
Number analyzed (Participants) | 67 | 64 | 68 | 64
Liters | 0.013 (0.025) | 0.171 (0.025) | 0.181 (0.025) | 0.163 (0.025)
Statistical Analysis 1: Comparison: Placebo vs UMEC 125 µg; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Covariance; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [0.088 to 0.229]
Statistical Analysis 2: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Covariance; Median Difference (Final Values) = 0.168, 95% CI 2-sided [0.099 to 0.238]
Statistical Analysis 3: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Covariance; Mean Difference (Final Values) = 0.150, 95% CI 2-sided [0.080 to 0.220]

2. Secondary Outcome: Change From Baseline in Weighted Mean 0-6 Hour FEV1 Obtained Post-dose at Day 1 and Day 28
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean FEV1 was derived by calculating the area under the FEV1/time curve (AUC), and then dividing the value by the time interval over which the AUC was calculated. The weighted mean was calculated using the 0-6 hour post-dose measurements at Days 1 and 28, which included pre-dose (30 minutes prior to dosing on Day 1, or 24 hours after the previous day's dose on Day 28), and post-dose at 15 minutes, 30 minutes, 1 hour, 3 hours, and 6 hours. Baseline is defined as the mean of the FEV1 values obtained at 30 minutes and immediately pre-dose on Day 1. Change from Baseline is defined as the difference between weighted mean at Days 1 and 28 and Baseline. Analysis was performed using a repeated measures model with covariates of Baseline, country, sex, age, treatment, smoking status, day, day by Baseline interaction, and day by treatment interaction.
Time Frame: Baseline, Day 1, and Day 28
Population: ITT Population. Participants (par.) with >=1 post-BL assessment and non-missing covariate data are included in the analysis. Different par. may have been analyzed at different time points (n=X, X, X, X in the category titles), so the overall number of par. analyzed reflects everyone in the ITT Population with data avaialable at >=1 time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 125 µg | UMEC 250 µg | UMEC 500 µg
Number analyzed (Participants) | 70 | 71 | 72 | 70
Liters
  Day 1, n=70, 70, 71, 70 | 0.005 (0.015) | 0.211 (0.015) | 0.224 (0.014) | 0.173 (0.015)
  Day 28, n=65, 64, 68, 64 | 0.009 (0.024) | 0.220 (0.024) | 0.204 (0.023) | 0.122 (0.024)

3. Secondary Outcome: Change From Baseline in Serial FEV1 Over 24 Hours After Dosing at Day 1 and Day 28
Description: Serial spirometry assessments were conducted on Day 1 and Day 28 over the course of 24 hours and were obtained 0 (Day 28 only), 1, 3, 6, 23, and 24 hours after dosing. Baseline is defined as the mean of the FEV1 values obtained at 30 minutes and immediately pre-dose on Day 1. Change from Baseline is defined as the difference between FEV1 on Days 1 and 28 and Baseline.
Time Frame: Baseline, Day 1, and Day 28
Population: ITT Population. All participants with >=1 post-BL assessment and non-missing covariate data are included in the analysis. Different participants may have been analyzed at different time points (represented by n=X, X, X, X in the category titles), so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 125 µg | UMEC 250 µg | UMEC 500 µg
Number analyzed (Participants) | 71 | 71 | 72 | 71
Liters
  Day 1, 1 hour, n=70, 71, 72, 71 | 0.013 (0.015) | 0.196 (0.015) | 0.212 (0.015) | 0.145 (0.015)
  Day 1, 3 hours, n=70, 71, 72, 71 | 0.008 (0.018) | 0.255 (0.018) | 0.274 (0.018) | 0.227 (0.018)
  Day 1, 6 hours, n=70, 71, 72, 70 | -0.004 (0.019) | 0.232 (0.019) | 0.221 (0.019) | 0.186 (0.019)
  Day 1, 23 hours, n=70, 70, 72, 70 | -0.036 (0.019) | 0.171 (0.019) | 0.186 (0.019) | 0.107 (0.019)
  Day 1, 24 hours, n=69, 71, 72, 70 | -0.002 (0.019) | 0.211 (0.018) | 0.216 (0.018) | 0.153 (0.018)
  Day 28, 0 hours, n=67, 64, 69, 65 | -0.017 (0.024) | 0.165 (0.024) | 0.203 (0.024) | 0.140 (0.024)
  Day 28, 1 hour, n=67, 64, 68, 65 | -0.008 (0.025) | 0.207 (0.026) | 0.182 (0.025) | 0.067 (0.026)
  Day 28, 3 hours, n=67, 65, 67, 64 | 0.008 (0.026) | 0.267 (0.026) | 0.204 (0.026) | 0.168 (0.026)
  Day 28, 6 hours, n=65, 65, 68, 64 | -0.005 (0.028) | 0.206 (0.028) | 0.181 (0.027) | 0.141 (0.028)
  Day 28, 23 hours, n=67, 64, 68, 64 | -0.013 (0.026) | 0.144 (0.027) | 0.161 (0.026) | 0.157 (0.027)
  Day 28, 24 hours, n=67, 64, 68, 64 | 0.024 (0.025) | 0.204 (0.026) | 0.192 (0.025) | 0.170 (0.026)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication up to 4 weeks.
Description: On-treatment serious adverse events (SAEs) and non-serious AEs are reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | Placebo | UMEC 125 µg | UMEC 250 µg | UMEC 500 µg
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/71 | 1/72 | 1/71
Other Adverse Events (participants affected / at risk) | 6/71 | 5/71 | 9/72 | 13/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | UMEC 125 µg (N=71) | UMEC 250 µg (N=72) | UMEC 500 µg (N=71)
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | UMEC 125 µg (N=71) | UMEC 250 µg (N=72) | UMEC 500 µg (N=71)
Headache (Nervous system disorders) | 3 | 3 | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6 | 8
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.